CLINICAL TRIAL: NCT02745535
Title: Safety, Tolerability and Efficacy of Sofosbuvir, Velpatasvir, and Voxilaprevir in Subjects With Previous DAA Experience
Acronym: RESOLVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Unity Health Care, Inc. (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Eleanor Wilson, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00067213
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C relapse
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOF/VEL/VOX (Experimental): Fixed dose combination of SOF/VEL/VOX (Sofosbuvir 400mg/Velpatasvir 100mg/ Voxilaprevir 100mg) dosed once daily for 12 weeks.
  Interventions: Drug: Sofosbuvir/Velpatasvir/Voxilaprevir

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir/Voxilaprevir
  Other Names: SOF/VEL/VOX; GS-7977/GS-5816/GS-9857

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) in adults with chronic hepatitis C infection who have failed to eradicate hepatitis C despite previous combination directly acting antiviral therapy.

DETAILED DESCRIPTION:
The treatment of chronic Hepatitis C with combination directly acting antiviral agents (DAAs) represents a dramatic improvement over previous therapies in safety, tolerability and efficacy, but these therapies are not universally effective. Some patients fail to achieve sustained virologic response (SVR) following therapy with combination DAAs, yet the ideal retreatment strategy for these patients has not yet been determined. As DAA medications become more widely available outside clinical trial settings, it is important to evaluate retreatment strategies in patients who fail combination DAA therapy, regardless of whether they had virologic failure, post-treatment relapse, or discontinued treatment prematurely.

The RESOLVE study will evaluate the safety, tolerability, and efficacy of treatment with a fixed dose combination of sofosbuvir (an approved NS5B inhibitor), velpatasvir (formerly GS-5816, a second generation NS5A inhibitor) and voxilaprevir (formerly GS-9857, an approved NS3/4A protease inhibitor) in HCV infected patients with early and advanced liver disease, including those with HIV or hepatitis B, who have failed previous combination DAA therapy. Patients with early stage and compensated cirrhosis will receive 12 weeks of therapy, and be followed for adverse events and SVR following completion of therapy.

RESOLVE will aid our understanding of the determinants of response to re-treatment with combination DAA therapy

* With and without cirrhosis
* In patients with HCV GT1 subtypes a and b
* In patients who previously failed DAA therapy
* With and without HIV or hepatitis B

RESOLVE will also examine factors associated with treatment response, including

* the viral and pharmacokinetics of patients receiving the combination of SOF/VEL/VOX, in patients with and without cirrhosis
* differential interferon sensitive gene responses
* host genetic and proteomic factors
* evolution of HCV quasispecies and resistance associated variants at baseline and in response to therapy
* changes in host HCV-specific immunity in patients with and without advanced liver disease

ELIGIBILITY:
Inclusion Criteria:

* Available for clinical follow-up through Week 44 after enrollment.
* Recurrent HCV GT-1
* Exposure to combination DAA therapy
* Able and willing to complete the informed consent process.
* Use of protocol specified methods of contraception
* Hepatitis B coinfected participants must have evidence of chronic infection and controlled on treatment
* HIV coinfected participants must have HIV status of one of the following:

  1. HIV untreated for >8 weeks prior to screening, CD4 >500, no intention of initiating ARV therapy for the duration of the trial.
  2. HIV suppressed on a stable, protocol-approved ARV regimen for >4 weeks prior to screening.

Exclusion Criteria:

* Combination DAA therapy was completed or discontinued less than 8 weeks prior to enrollment.
* Current or prior history of any clinically significant illness, organ transplantation, and/or concomitant medication that may interfere with the subject treatment, assessment of compliance with the protocol.
* Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency, cholangitis)
* Laboratory results outside acceptable ranges at screening.
* Female who is pregnant, breast-feeding or planning to become pregnant during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Wilson, MD, Principal Investigator — University of Maryland Institute of Virology
Locations (1):
- Institute of Human Virology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment opened 5-May-2016 and closed 24-Jan-2018. All study visits were done in an outpatient medical clinic in Baltimore or Washington DC.
Pre-assignment Details: Participants infected with chronic hepatitis C (HCV), genotype 1, who previously were treated with unsuccessful combination DAA-based therapy were enrolled in the study. Subjects included HCV mono-infection, HCV/HIV co-infection or HCV/hepatitis B (HBV) co-infection or HCV/HIV/HBV triple-infected patients.
Groups:
- SOF/VEL/VOX: Fixed dose combination of SOF/VEL/VOX (Sofosbuvir 400mg/Velpatasvir 100mg/ Voxilaprevir 100mg) dosed once daily for 12 weeks in participants with chronic hepatitis c previously exposed to direct acting antivirals (DAA).
Period: Overall Study
Arm/Group | SOF/VEL/VOX
Started | 77
Sustained Virologic Repsonse | 70 (Sustained Virologic response measured 24 weeks after completing study medication)
Completed | 71 (Completed 12 weeks of study medication per protocol)
Not Completed | 6
Not completed — Death | 1
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Participants with compensated cirrhosis and non cirrhotic were enrolled. Participants co-infected with HIV ( as well as triple infected with HIV, hepatitis B and hepatitis C were included in the study.
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 76
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 66
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 77
Compensated cirrhotic [Count of Participants; unit: Participants] | 31
Co-infected with HIV [Count of Participants; unit: Participants] | 22
Coinfected with HIV and hepatitis B [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 and 4 Adverse Events
Description: Number of participants with grade 3 and 4 adverse events during treatment with and/or within 30 of completion of SOF/VEL/VOX in HCV infected
Time Frame: up to 16 weeks
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 77
Participants | 12

2. Primary Outcome: Number of Participants Who Achieve Sustained Virologic Response (SVR) 12 Weeks After Completion of Therapy (SVR12)
Description: Intention to treat (ITT) analysis. Sustained Virologic Response as measure by an undetectable HCV RNA level 12 weeks after completion of therapy.
Time Frame: Post-treatment week 12
Population: All participants who took at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 77
Participants | 70

3. Secondary Outcome: Number of Participants Who Achieve End of Treatment Virologic Response (ETR) at Completion of Therapy.
Description: Per protocol analysis. End of Treatment Virologic Response as measure by an undetectable HCV RNA level completion of therapy.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 71
Participants | 71

4. Secondary Outcome: Number of Participants Who Achieve Sustained Virologic Response (SVR) 4 Weeks After Completion of Therapy.
Description: Per protocol analysis. Sustained Virologic Response as measure by an undetectable HCV RNA level 4 weeks after completion of therapy.
Time Frame: Post-treatment week 4
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 71
Participants | 70

5. Secondary Outcome: Number of Participants Who Achieve Sustained Virologic Response (SVR) 24 Weeks After Completion of Therapy.
Description: Per protocol analysis. Sustained Virologic Response as measure by an undetectable HCV RNA level 24 weeks after completion of therapy.
Time Frame: Post-treatment week 24
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL/VOX
Number analyzed (Participants) | 71
Participants | 70

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and reported from day first dose of study medication was taken until 30 days after last dose, which was an average of 16 weeks.
Description: \Participants were assessed for adverse events at every follow up visit. Adverse events were monitored from the time of informed consent until last study visit.
Arm/Group | SOF/VEL/VOX
All-Cause Mortality (participants affected / at risk) | 1/77
Serious Adverse Events (participants affected / at risk) | 12/77
Other Adverse Events (participants affected / at risk) | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOF/VEL/VOX (N=77)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypertensive stroke (Vascular disorders) | 1 (1)
Pulmonary hypertension, exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subderal hematoma, traumatic (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase >5xULN (Investigations) | 1 (1)
Creatinine >2x baseline (Investigations) | 2 (2)
Glucose level >250mg/dL (Investigations) | 2 (2)
INR >2x ULN (Investigations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOF/VEL/VOX (N=77)
Fatigue (General disorders) | 21 (21)
Headache (Nervous system disorders) | 19 (19)
Diarrhea (Gastrointestinal disorders) | 16 (16)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT02745535/Prot_SAP_000.pdf